CLINICAL TRIAL: NCT02583321
Title: Detection of Chlorhexidine in Tracheal Secretions After Routine Oral Care With Chlorhexidine Gluconate: an Ancillary Study of the DEMETER Trial (NCT02515617)
Brief Title: Detection of Chlorhexidine in Tracheal Secretions After Routine Oral Care With Chlorhexidine Gluconate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Collaborators: Ministry of Health, France (Other Government); University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CHD 054-15
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Chlorhexidine; Intensive Care
Keywords: chlorhexidine gluconate; oral care; mechanical ventilation; critically ill patients; tracheal secretions; subglottic secretions

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Period with endotracheal tubes not allowing SSD (Active Comparator): During this period of the DEMETER study (NCT02515617), patients will be intubated with standard endotracheal tubes not allowing Subglottic Secretions
  Interventions: Device: Endotracheal tubes not allowing SSD
- Period with endotracheal tubes allowing SSD (Experimental): During this period of the DEMETER study (NCT02515617), patients will be intubated with specific endotracheal tubes allowing Subglottic Secretions Drainage
  Interventions: Device: Endotracheal tubes allowing SSD

INTERVENTIONS:
Device: Endotracheal tubes not allowing SSD — In the participating center, a bundle of Ventilator-Associated Pneumonia (VAP) prevention will be applied: elevate the head of the bed to 30°-45°, regular oral care, manage patients with sedation algorithm, assess readiness to extubate daily, intermittent control of endotracheal tube cuff pressure
  Arms: Period with endotracheal tubes not allowing SSD
Device: Endotracheal tubes allowing SSD — In the participating center, a bundle of VAP prevention will be applied: elevate the head of the bed to 30°-45°, regular oral care, manage patients with sedation algorithm, assess readiness to extubate daily, intermittent control of endotracheal tube cuff pressure.
  In addition, SSD will be realized using a 10 ml syringe at in attending frequency of 2 hours.
  Arms: Period with endotracheal tubes allowing SSD

SUMMARY:
Recent meta-analysis have suggested that the safety of oral care with chlorhexidine in patients under mechanical ventilation could be questionable. Whatever the hypothetical mechanisms involved (direct cellular toxicity, underdiagnosis of Ventilator-Associated Pneumonia), presence of chlorhexidine in tracheal secretions after routine oral care is the cornerstone of this potential side effect of the routine oral care with chlorhexidine gluconate. The DEMETER study assessing the medico-economical impact of the subglottic secretions drainage study (NCT02515617) provides the opportunity to perform this proof of concept study (detection of chlorhexidine in tracheal secretions after routine oral care with chlorhexidine gluconate) and to evaluate the impact of the subglottic secretion drainage on this potential detection of chlorhexidine.

This ancillary study will be performed in one of the centers participating to the DEMETER study.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Invasive mechanical ventilation (MV) delivered via an endotracheal tube and MV required more than 72 hours
* Intubation performed in units in which the specific endotracheal tube allowing the subglottic secretions drainage (SSD) will be available during the SSD period of the trial
* Information delivered

Exclusion Criteria:

* Previous inclusion in the study
* Patients moribund at the ICU admission
* Pregnant, parturient or breast-feeding woman
* Patient hospitalized without consent and/or deprived of liberty by court's decision
* Patient under guardianship or curators
* Lack of social insurance
* Concomitant inclusion in a trial on VAP prevention
* Patient with no comprehension of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
Rate of patients with detection of chlorhexidine in tracheal secretions during the period without SSD | Day 3 of mechanical ventilation

SECONDARY OUTCOMES:
Rate of patients with detection of chlorhexidine in tracheal secretions during the period with SSD | Day 3 of mechanical ventilation
Cumulative incidence of detection of chlorhexidine in tracheal secretions according to the study group. | Day 28 of mechanical ventilation
Rate of patients with detection of chlorhexidine in subglottic secretions during the period with SSD | Day 3 of mechanical ventilation
Cumulative incidence of detection of chlorhexidine in subglottic secretions during the SSD period. | Day 28 of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude LACHERADE, MD, Principal Investigator — CHD VENDEE; Bertrand Diquet, Ph.D, Principal Investigator — University Hospital, Angers
Locations (1):
- CHD Vendee, La Roche-sur-Yon, France

REFERENCES:
- [Background] Klompas M, Speck K, Howell MD, Greene LR, Berenholtz SM. Reappraisal of routine oral care with chlorhexidine gluconate for patients receiving mechanical ventilation: systematic review and meta-analysis. JAMA Intern Med. 2014 May;174(5):751-61. doi: 10.1001/jamainternmed.2014.359. PMID 24663255
- [Background] Price R, MacLennan G, Glen J; SuDDICU Collaboration. Selective digestive or oropharyngeal decontamination and topical oropharyngeal chlorhexidine for prevention of death in general intensive care: systematic review and network meta-analysis. BMJ. 2014 Mar 31;348:g2197. doi: 10.1136/bmj.g2197. PMID 24687313